CLINICAL TRIAL: NCT00612755
Title: Open, Randomized, Multicenter Phase IV Study to Evaluate Efficacy and Safety to Extend Treatment 24 Weeks in co-Infected HIV-HCV Patients Genotype 1 and/or 4
Brief Title: Efficacy and Safety to Extend Treatment 24 Weeks in co-Infected HIV-HCV Genotype 1 and/or 4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinico Universitario San Cecilio (Other)
Responsible Party: José Hernández-Quero, Hospital Clinico Universitario San Cecilio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Extrados; 2004-004948-45
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: HIV Infections; Hepatitis C
Keywords: chronic hepatitis C; co-infection; extend treatment; co-infected HIV-HCV
MeSH Terms: conditions — HIV Infections; Hepatitis C; Hepatitis C, Chronic; Coinfection | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Peginterferon alfa-2a 180 mcg/week + 1000-1200 mg/day ribavirin during 24 weeks
  Interventions: Drug: Peginterferon alfa-2a + ribavirin
- 2 (No Intervention)

INTERVENTIONS:
Drug: Peginterferon alfa-2a + ribavirin — Peginterferon alfa-2a 180 mcg/week ribavirin 1000-1200 mg/day during 24 weeks
  Other Names: Pegasys
  Arms: 1

SUMMARY:
A study concerning viral kinetic with 10 co-infected HIV-HCV patients on treatment with peginterferon alfa-2a + ribavirin o IFN + ribavirin was reported in Conference on Retroviruses and Opportunistic Infections 2002 by Dr. Torriani shown half-life of HCV virions and the viral clearance was larger than mono-infected patients.

The doubt is if this difference in viral kinetic of HIV-HCV co-infected patients versus mono-infected is related with the loss of profited on treatment.

In the APRICOT trial patients genotype 2/3 were treated for 48 weeks and the relapse rates was only 2%.

The present study want to evaluate is the treatment extent for 24 weeks more in patients genotype 1 and/or 4 will be improve the percentage of patients with viral clearance at the end of the follow-up period, to prevent relapsed in patients with response at the end of treatment.

Patients will be randomized to received 180 µg/week of peginterferon alfa-2a + 1000-1200 mg/day of ribavirin during 24 weeks more or control.

DETAILED DESCRIPTION:
To evaluate efficacy of extend treatment during 24 weeks more in co-infected HIV-HCV patients with genotype 1 and/or 4 who at 44 week of treatment with peginterferón alfa-2a in combination with ribavirin have RNA-HCV undetectable.

ELIGIBILITY:
Inclusion Criteria:

* Patients on treatment with Peginterferon alfa-2a (180 µg/week) in combination with Ribavirin (1000-1200 mg/day) who are RNA-HCV undetectable at 44 week
* RNA-HCV positive at 48 week before study and genotype 1 or 4.
* HIV-1 positive: ELISA y Western-blot.
* Stable status of HIV-1 infection in the opinion of the investigator, (patients who are not expected to progress during the study).
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug. Additionally, all fertile males and females must be using two forms of effective contraception during treatment and during the 6 months after treatment end. This may include, but is not limited to, using birth control pills, IUDs, condoms, diaphragms, or implants, being surgically sterilized, or being in a post-menopausal state.
* Willingness to give written informed consent and willingness to participate to and comply with the study.

Exclusion Criteria:

* Patients with RNA-HCV detectable after 44 weeks of treatment with Peginterferon alfa-2a (180 µg/week) in combination with Ribavirin (1000-1200 mg/day).
* Patients with other treatment for chronic hepatitis, different which of inclusion criteria is described.
* More of tree weeks from the end of treatment with Peginterferon alfa-2a (180 µg/week) in combination with Ribavirin (1000-1200 mg/day) to the inclusion in "EXTRADOS" trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
% of patients with RNA-HCV undetectable | at 48 week of study (24 weeks after the end of treatment period of trial).

SECONDARY OUTCOMES:
% of percentage of patients with RNA-HCV undetectable | 24 weeks of trial period

CONTACTS AND LOCATIONS:
Overall Officials: José Hernández-Quero, Dr, Study Chair — Hospital Clínico Universitario San Cecilio
Locations (19):
- Spain (19):
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Insular, Las Palmas, Gran Canaria
  - Hospital Clínico Universitario San Cecilio, Granada, Granada
  - Hospital de Donostia, San Sebastián, Guipúzcoa
  - Complejo Hospitalario Universitario, Santiago, La Coruña
  - Fundación Hospital de Alcorcón, Alcorcón, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Son Dureta, Palma de Mallorca, Mallorca
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital de Valme, Seville, Sevilla
  - Consorcio Hospital General, Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid, Valladolid